CLINICAL TRIAL: NCT01823783
Title: Endomysial Fibrosis, Muscular Inflammatory Response and Calcium Homeostasis Dysfunction : Potential Links and Targeted Pharmacotherapy in Duchenne Muscular Dystrophy (DMD).
Brief Title: Endomysial Fibrosis, Muscular Inflammatory Response and Calcium Homeostasis Dysfunction in Duchenne Muscular Dystrophy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8948
Record Dates: First submitted 2013-03-22; First posted 2013-04-04 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Duchenne Muscular Distrophy (DMD)
Keywords: Duchenne muscular distrophy; Endomysial Fibrosis; Muscular Inflammatory Response; Calcium Homeostasis Dysfunction; Muscle biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DMD infant (Other): Muscle biopsy
  Interventions: Other: Muscle biopsy
- Control infant (Other): Muscle biopsy (during lower limb operation surgery for pure orthopedic causes)
  Interventions: Other: Muscle biopsy

INTERVENTIONS:
Other: Muscle biopsy — Muscle biopsy

SUMMARY:
Duchenne muscular dystrophy (DMD) is the most common and devastating form of muscular dystrophy, caused by an X-chromosome gene mutation resulting in the absence of the protein dystrophin. Gene therapy by exon skipping or stop codon read-through and cell therapy are at the stage of clinical assays with very promising results. Nevertheless, they will not allow a complete cure of DMD patients and they will concern only specific types of mutations. It is therefore crucial to develop other therapeutic strategies related to the natural history of the disease and targeted not on the dystrophin itself, but on the consequences of its absence.

Another crucial pathophysiological pathway in DMD is muscle cell calcium homeostasis, particularly via the ryanodine recepteur (RyR1).

Our study focus on the relationship between endomysial fibrosis, abnormal inflammation response and calcium homeostasis dysfunction which are not entirely established in DMD.

The identification of the biological mechanisms that play a role in the severity of the phenotype, particularly endomysial fibrosis, should allow the development of targeted pharmacotherapy as a complementary strategy for the future treatment of DMD.

ELIGIBILITY:
Inclusion Criteria:

* Boy between 2 to 15 years old.
* Lack of any infectious disease in the last week before the study.
* Consent form signed by parents.

Inclusion Criteria for DMD infant

* Clinical suspicion of Duchenne Muscular Dystrophy

Inclusion Criteria for Control healthy Infant

* Lack of any antecedent of congenital cardiac, pulmonary or muscular disease including DMD.

Exclusion Criteria:

* Subjects who are unable or unwilling to tolerate study constraints
* Parents of the subject unable or unwilling to undergo informed consent
* Subject with no rights from the national health insurance programme

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2012-11-07 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Quantification of endomysial fibrosis | 1 day (biopsy day)
quantification of the muscle inflammation | 1 day (biopsy day)
  * Measure of the protein (Immunofluorescence and western blot) and mRNA (qRT-PCR) expression of the following markers of muscular inflammation response
  * Presence and quantification of cellular partners of inflammation and muscle regeneration (M1 (CD68/KP1) and M2 (CD206) macrophages, quiescent and activated satellite cells (CD56/NCAM) and endothelial cells (CD31/PECAM-1)).

CONTACTS AND LOCATIONS:
Overall Officials: François RIVIER, PU PH, Principal Investigator — uh montpellier
Locations (7):
- France (7):
  - UH Bordeaux, Bordeaux
  - UH Lille, Lille
  - Montpellier University Hospital, Montpellier
  - Necker Hospital, Paris
  - UH Reims, Reims
  - UH Saint Etienne, Saint-Etienne
  - UH Toulouse, Toulouse